CLINICAL TRIAL: NCT06552442
Title: Intracoronary Administration of Glucocorticoids as a Treatment Method for No-Reflow Phenomenon in STEMI Patients
Brief Title: Intracoronary Administration of Glucocorticoids as a Treatment Method for No-Glucocorticoid Treatment for No-Reflow in STEMI
Acronym: GCT-NR-STEMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amosov National Institute of Cardiovascular Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ethics Protocol Number 1/2020
Record Dates: First submitted 2024-07-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Ischemia-reperfusion Injury; No-reflow
Keywords: acute coronary syndrome; STEMI; No-reflow; Intracoronary; Glucocorticoids
MeSH Terms: conditions — Reperfusion Injury; Acute Coronary Syndrome; ST Elevation Myocardial Infarction | interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: The main study group receives intracoronary methylprednisolone for the no-reflow phenomenon. The control group does not receive any pharmacological intervention. Considering that this complication is very rare, the control group was selected retrospectively.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Main group (Experimental): Main group - 10 patients. STEMI patients with the occurrence of the no-reflow phenomenon after stenting of the infarct-related artery.
  Treatment of the phenomenon: intracoronary administration of methylprednisolone.
  Interventions: Drug: Methylprednisolone
- Control group (No Intervention): Control group - 10 patients. STEMI patients with the occurrence of the no-reflow phenomenon after stenting of the infarct-related artery.
  Treatment of the phenomenon: no pharmacological intervention.

INTERVENTIONS:
Drug: Methylprednisolone — High-dose intracoronary glucocorticoid methylprednisolone to abrogate no-reflow: a unique study for restoration of infarct-related artery patency and reduction of ischemia-reperfusion injury
  Arms: Main group

SUMMARY:
The goal of this clinical trial is to improve reperfusion therapy in STEMI patients with no-reflow phenomenon. Based on literature review and pathological studies, the investigators believe that myocardial ischemia-reperfusion injury is primarily due to myocardial edema, which is angiographically manifested by the no-reflow. To restore blood flow, high-dose intracoronary methylprednisolone was applied. The main idea is to stabilize cell membranes and stop the progression of edema. It is local, not systemic, single administration that avoids serious side effects. The primary hypothesis is that hormone administration will improve blood flow to TIMI 2/3 in TIMI 0/1after stenting infarct-related artery.

DETAILED DESCRIPTION:
The study involves comparing the main group receiving intracoronary methylprednisolone with a group of patients without intracoronary pharmacotherapy. Preliminary results: the use of methylprednisolone allows for the restoration of coronary blood flow but does not affect mortality.

ELIGIBILITY:
Inclusion Criteria:

* TIMI 0/1 flow after successful artery obstruction stenting
* Men and women aged 40 years and older

Exclusion Criteria:

* Coronary artery dissection
* Abrupt intraoperative coronary artery closure
* Intraoperative thrombosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Restoration of coronary blood flow | 3 minutes
  Degree of restoration of coronary blood flow on the Thrombolysis in myocardial infarction (ТIMI) grade 0-3 (3 is the best result, 0/1 - bad or no-reflow) from TIMI 0 or TIMI 1 to TIMI 2 or TIMI 3

CONTACTS AND LOCATIONS:
Locations (1):
- Amosov National Institute of cardiovascular surgery, Kyiv, Amosov Street, 6, Ukraine